CLINICAL TRIAL: NCT02750033
Title: Intraoperative Margin Assessment During Mohs Surgery
Status: Withdrawn | Type: Observational
Why Stopped: Protocol changed to meet IRB requirements for patient safety
Sponsor: Seton Healthcare Family (Other)
Collaborators: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Jason Reichenberg, MD, Seton Healthcare Family
Other Study IDs: CR-16-049
Record Dates: First submitted 2016-04-20; First posted 2016-04-25 (Estimated); Last update posted 2018-08-20 (Actual); Status verified 2018-08

CONDITIONS: Squamous Cell Carcinoma (SCC); Basal Cell Carcinoma (BCC)
MeSH Terms: conditions — Carcinoma, Squamous Cell; Carcinoma, Basal Cell

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Basal Cell Carcinoma (BCC): Adult patients undergoing Mohs surgery to remove basal cell carcinoma (BCC) will have surgical margins assessed with multimodal optical spectroscopy (MMS) device, as well as standard histopathology evaluation.
  Interventions: Device: Multimodal Spectroscopy (MMS)
- Squamous Cell Carcinoma (SCC): Adult patients undergoing Mohs surgery to remove squamous cell carcinoma (BCC) will have surgical margins assessed with multimodal optical spectroscopy (MMS) device, as well as standard histopathology evaluation.
  Interventions: Device: Multimodal Spectroscopy (MMS)

INTERVENTIONS:
Device: Multimodal Spectroscopy (MMS) — surgical margin assessment with multimodal optical spectroscopy (MMS) device

SUMMARY:
The research team will develop an intraoperative handheld device for assessing surgical margins during Mohs surgery. The device technology is based on multimodal optical spectroscopy (MMS), combining three optical spectroscopy techniques into one device. The researchers will first acquire proof of concept MMS measurements within the Mohs surgery suite immediately after surgical excision and prior to histological processing. MMS measurements will be acquired directly on the patient from the NMSC excision site. The final outcome of this study will result in the sensitivity and specificity of MMS compared to histopathology during Mohs surgery. These results will allow for the estimation of the potential benefit of an intraoperative margin assessment technique.

DETAILED DESCRIPTION:
Acquire intraoperative MMS measurements in vivo. After assessing this approach on excised tissues, MMS measurements will be aquired directly on the patient from the NMSC excision site. MMS data will be acquired on patients being treated for NMSC at the Austin Dermatologic Surgery Center, the surgical site for the dermatology practice of Seton/University of Texas Physicians group. Similar to the measurements on freshly excised tissues, MMS data will be acquired in a grid pattern on the excision site. The site will be blotted with gauze to remove residual blood prior to the measurement, and continuously blotted as needed until all measurements have been taken. The handheld probe of the MMS enables assessment of both the wound periphery and deeper layers of tissue to determine if any tumor is remaining. For this initial pilot study, we plan to take measurements on 10 patients (5 BCC, 5 SCC), along with corresponding normal tissue measurements.

Retrospective analysis of MMS sensitivity and specificity. The MMS technique is an information rich modality providing both morphological and functional parameters of the interrogated tissue that could be correlated to known tumor pathology. However, this extracted information will require development of sophisticated spectral analysis models which would be beyond the scope of the current study. Therefore, for the purpose of this study, standard statistical techniques will be used to determine the classification power of MMS for tumor margin detection. While this approach does not fully elucidate the underlying pathology responsible for the classification, these types of models have been shown to perform at or better than those based on a morphological approach. This approach has been previously employed to classify skin cancer with high diagnostic accuracy. The final outcome of this study will result in the sensitivity and specificity of MMS compared to histopathology during Mohs surgery. These results will allow for the estimation of the potential benefit of an intraoperative margin assessment technique. This type of retrospective study will provide a proof of concept that would warrant further development and prospective studies of the MMS approach.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female and over 18 years of age.
2. Patients undergoing Mohs surgery for SCC or BCC

Exclusion Criteria:

1. Male or Female and under 18 years of age.
2. Patients with diagnosis other than SCC or BCC

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing Mohs surgery to remove basal or squamous cell carcinoma.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity of MMS compared to histopathology during Mohs surgery | May, 2016 to December, 2016 up to 6 moths

CONTACTS AND LOCATIONS:
Overall Officials: Jason Reichenberg, MD, Principal Investigator — Seton Healthcare Family

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Robinson JK. Sun exposure, sun protection, and vitamin D. JAMA. 2005 Sep 28;294(12):1541-3. doi: 10.1001/jama.294.12.1541. No abstract available. PMID 16193624
- [Background] Asgari MM, Olson JM, Alam M. Needs assessment for Mohs micrographic surgery. Dermatol Clin. 2012 Jan;30(1):167-75, x. doi: 10.1016/j.det.2011.08.010. PMID 22117877
- [Background] Koslosky CL, El Tal AK, Workman B, Tamim H, Durance MC, Mehregan DA. Reliability of skin biopsies in determining accurate tumor margins: a retrospective study after Mohs micrographic surgery. Dermatol Surg. 2014 Sep;40(9):964-70. doi: 10.1097/01.DSS.0000452621.79017.19. PMID 25099294
- [Background] Sharma M, Marple E, Reichenberg J, Tunnell JW. Design and characterization of a novel multimodal fiber-optic probe and spectroscopy system for skin cancer applications. Rev Sci Instrum. 2014 Aug;85(8):083101. doi: 10.1063/1.4890199. PMID 25173240
- [Background] Lim L, Nichols B, Migden MR, Rajaram N, Reichenberg JS, Markey MK, Ross MI, Tunnell JW. Clinical study of noninvasive in vivo melanoma and nonmelanoma skin cancers using multimodal spectral diagnosis. J Biomed Opt. 2014;19(11):117003. doi: 10.1117/1.JBO.19.11.117003. PMID 25375350